CLINICAL TRIAL: NCT00624754
Title: recipientsProspective Evaluation of the Efficacy of Budesonide/Formoterol (Symbicort®) in Bronchiolitis Obliterans in Allogeneic Haematopoietic Stem Cell Transplantation (AHSCT) Recipients
Brief Title: Prospective Evaluation of the Efficacy of Budesonide/Formoterol in Bronchiolitis Obliterans in AHSCT
Acronym: Alloforb
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P070116
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2009-01

CONDITIONS: Obstructive Airway Disease
Keywords: Obstructive airway disease; bronchiolitis obliterans; allogeneic hematopoietic stem cell transplantation; bone marrow transplantation; inhaled treatment; Budesonide Formoterol
MeSH Terms: conditions — Lung Diseases, Obstructive; Bronchiolitis Obliterans | interventions — Formoterol Fumarate; Budesonide; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients with OAD will receive Symbicort® at the dose of two puffs morning and evening, each delivering 400/12 µg of budesonide/formoterol. Symbicort® will be administered by inhalation using the Turbuhaler (TH) system
  Interventions: Drug: Formoterol/Budesonide
- 2 (Placebo Comparator): Patients with OAD will receive lactose as a placebo, administered by inhalation using the Turbuhaler (TH) system
  Interventions: Drug: lactose

INTERVENTIONS:
Drug: Formoterol/Budesonide — Budesonide/Formoterol 400/12: 800 µg b.i.d for 1 month
  Arms: 1
Drug: lactose — Lactose 2 puffs b.i.d for 1 month
  Arms: 2

SUMMARY:
The usual treatment for obstructive airway disease (OAD) after allogeneic hematopoietic stem cell transplantation (AHSCT) , which is related to graft versus host disease (GVHD), consists of intensification of systemic immunosuppressive therapy.

DETAILED DESCRIPTION:
Although it has not been evaluated prospectively, the usual treatment for obstructive airway disease (OAD) after allogeneic hematopoietic stem cell transplantation (AHSCT) , which is related to graft versus host disease (GVHD), consists of intensification of systemic immunosuppressive therapy. However, this treatment has a limited efficacy and is associated with a significant number of serious adverse effects, particularly infectious. Alternative treatments are therefore necessary.We have retrospectively reported clinical and functional improvement in patients with OAD following AHSCT treated with inhaled budesonide/formoterol combination.These encouraging results need to be confirmed by the present randomised, prospective double-blind trial. This study is therefore designed to evaluate the efficacy of budesonide/formoterol versus placebo in patients with moderate to severe OAD, not requiring initiation or intensification of systemic immunosuppressive therapy for extra thoracic GVHD.

Inclusion criteria modified according to amendment of 02/11/2009

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years.
* Previous normal PFTs available.
* Absence of extrathoracic GVH disease justifying initiation or intensification of systemic immunosuppressive therapy.
* Respiratory signs present for less than 6 months.
* AHSCT recipients who have developed moderate to severe bronchiolitis obliterans, defined by reduction of FEV1/VC below the 5th percentile of predicted normal or < 80% of predicted, with FEV1 < 80% of predicted and ≥ 40% of predicted, not reversible after inhalation of short-acting beta-2 agonist. AHSCT recipients with FEV1 < 80% of predicted and ≥ 40% of predicted, not reversible after inhalation of short-acting beta-2 agonist and TLC ≥ 80% of predicted.
* Respiratory symptoms related to obstructive lung disease present for at least 6 months.
* Negative respiratory microbiology work-up.
* Informed consent signed by the patient or both parents of a minor.

Exclusion Criteria:

* Extrathoracic graft versus host reaction justifying initiation or intensification of systemic immunosuppressive therapy.
* Use of inhaled bronchodilator and/or corticosteroid therapy at the time of inclusion.
* Known intolerance to inhaled bronchodilators and/or corticosteroids and/or lactose.
* Personal or donor history of asthma.
* Active smoking
* FEV1 < 40% of predicted normal or ≥ 80% of predicted normal or PO2 < 50 mmHg.
* Documented respiratory tract infection.
* Pregnancy.
* Absence of effective contraception during the trial.
* Not covered by French national health insurance.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is based on pulmonary function tests (PFT): the absolute variation of FEV1 after 1 month of treatment will be assessed. | 1 month

SECONDARY OUTCOMES:
Improvement or stabilisation of FEV1; Prevalence of improvement of FEV1 by at least 200 ml and 12% at 1 month compared to baseline; Variation of FEF 25-75% and vital capacity; Quality of life measurement; Evaluation of the clinical score | 1, 6 and 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne BERGERON, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Saint Louis, Paris, France

REFERENCES:
- [Background] Bergeron A, Belle A, Chevret S, Ribaud P, Devergie A, Esperou H, Ades L, Gluckman E, Socie G, Tazi A. Combined inhaled steroids and bronchodilatators in obstructive airway disease after allogeneic stem cell transplantation. Bone Marrow Transplant. 2007 May;39(9):547-53. doi: 10.1038/sj.bmt.1705637. Epub 2007 Mar 12. PMID 17351647
- [Derived] Bergeron A, Chevret S, Chagnon K, Godet C, Bergot E, Peffault de Latour R, Dominique S, de Revel T, Juvin K, Maillard N, Reman O, Contentin N, Robin M, Buzyn A, Socie G, Tazi A. Budesonide/Formoterol for bronchiolitis obliterans after hematopoietic stem cell transplantation. Am J Respir Crit Care Med. 2015 Jun 1;191(11):1242-9. doi: 10.1164/rccm.201410-1818OC. PMID 25835160